CLINICAL TRIAL: NCT01476683
Title: An Open-Label, Fasting, Crossover, Single-Dose Pharmacokinetic Study of Four Formulations of Racecadotril
Brief Title: Study to Compare the Pharmacokinetics Profiles of Four Racecadotril Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: RACDIR1002
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Diarrhea
Keywords: Antidiarrheals
MeSH Terms: conditions — Diarrhea | interventions — racecadotril

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- FCT (Experimental): A single 2 x100 mg dose of an experimental Racecadotril Film-coated tablet (FCT) administered orally with 240 ml of water, with a 7- day washout between visits.
  Interventions: Drug: Racecadotril
- RPB (Experimental): A single 2 x100 mg dose of an experimental Racecadotril Powder Blend administered orally with 240 ml of water, with a 7- day washout between visits.
  Interventions: Drug: Racecadotril
- TFT (Active Comparator): A single 2 x 100 mg dose of a marketed Tiorfast® capsule administered orally with 240 ml of water, with a 7-day washout between visits.
  Interventions: Drug: Racecadotril
- TFR (Active Comparator): A single 175 mg dose of a marketed Tiorfanor® 175 mg FCT administered orally with 240 ml of water, with a 7-day washout between visits.
  Interventions: Drug: Racecadotril

INTERVENTIONS:
Drug: Racecadotril — Film-coated tablet
  Other Names: Not yet marketed
  Arms: FCT
Drug: Racecadotril — Racecadotril Powder Blend
  Other Names: Not yet marketed
  Arms: RPB
Drug: Racecadotril — Marketed Capsule
  Other Names: Tiorfast®
  Arms: TFT
Drug: Racecadotril — Marketed Film-coated Tablet
  Other Names: Tiorfanor®
  Arms: TFR

SUMMARY:
This study is designed to compare the pharmacokinetics of four products used for treatment of acute diarrhea.

DETAILED DESCRIPTION:
The study will be a single dose, randomized, four -way, four-sequence crossover study in 24 healthy subjects, with equal numbers of males and females (minimum of 10 of either gender). Subjects who drop out will not be replaced. The four doses of medication given in the study (a single dose in each of the four study periods) will be separated by a washout period of at least 7 calendar days. In each study period, 17 blood samples for pharmacokinetic analysis will be taken over 12 hours. Blood samples will be centrifuged and concentrations of thiorphan (the active metabolite) in plasma will be measured using a validated chromatographic assay. Pharmacokinetic parameters will be calculated from plasma concentration data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects (equal numbers of males and females)
* Volunteers aged of at least 18 years but not older than 55 years
* Subjects will have a Body Mass Index (BMI) within protocol-specified parameters.
* Non- or ex-smokers; an ex-smoker being defined as someone who completely stopped smoking for at least 12 months before day 1 of this study.
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations Has signed and dated the informed consent document, indicating that the subject has been informed of all pertinent aspects of the study
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Seated pulse rate and blood pressure within protocol-specified parameters.
* Relationship to persons involved directly with the conduct of the study (i.e., principal investigator; sub-investigators; study coordinators; other study personnel; employees or contractors of the sponsor or Johnson & Johnson subsidiaries; and the families of each)
* Females who are pregnant or are lactating
* Females of childbearing potential or males with a female partner of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the entire duration of the study
* History of significant hypersensitivity to racecadotril or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Use of certain drugs/medications within protocol-specified timeframes
* Medical history or condition that may, per protocol or in the opinion of the investigator, adversely affect the safety of the study subject or compromise study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration | Pre-dose and 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10 and 12 hours post drug administration
  Maximum Observed Plasma Concentration (Cmax), which is the maximum (peak) concentration (amount of drug) measurable in blood plasma after a dose is administered, measured in nanograms/milliliter (ng/mL)
AUC(0-t) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10 and 12 hours post drug administration
  AUC(0-t) is the area under the plasma concentration verses time curve from start of drug administration until the time of the last measurable plasma concentration, calculated as hour*nanograms (ng) per milliliter (mL).
AUC(0-∞) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10 and 12 hours post drug administration
  AUC (0-∞) is the area under the plasma concentration-vs.-time curve from start of drug administration until infinity.

SECONDARY OUTCOMES:
Time of Maximum Concentration | During 12 hours post-dose
  The time at which maximum concentration is reached (Tmax)
Terminal Elimination Rate Constant | During 12 hours post-dose
  The Terminal Elimination Rate Constant (Lamda z) is the time required to eliminate half the administered dose
Terminal Phase Plasma Half-Life | During 12 hours post-dose
  Terminal phase plasma half-life (t ½) is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, rather than the time required to eliminate half the administered dose.
Lag Time | During 12 hours post-dose
  The time delay between drug administration and the quantification of absorption

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada